CLINICAL TRIAL: NCT07080723
Title: Algorithm Guided Treatment Versus Treatment as Usual (TAU) for Patients With Treatment Resistant Depression
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, René Ernst Nielsen, Clinical Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20250007
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: Algorithm guided treatment; AGT; ALGO; Treatment as usual; TAU; Treatment resistant depression; TRD; Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm guided treatment (AGT) (Experimental): Treatment choice is defined in the AGT group by predetermined steps and critical decision points. The critical decision point moment is predetermined and marks the patient's outpatient visit. At these timepoint, HAMD score is determined and change from last visit is calculated, and based on this evaluation, specific treatment revisions are made following established "if-then" decision rules. This implies that the subsequent step is determined by the outcome of the assessment. If the patient's condition is assessed satisfactory, one step is selected and if the desired outcome is not achieved, an alternative step is pursued. Treatment choice for each step is based on patients medical history, previous therapy effect, adverse events, evidence based medicine and is selected a priori when patients are randomized by discussion with a senior consultant. AGT consists of which treatments to use at each step, how to implement each treatment and in what order to implement different treatments.
  Interventions: Other: Algorithm guided treatment (AGT)
- Treatment as usual (TAU) (Active Comparator): TAU group treatment is defined and supervised by senior consultants with an experience in a treatment of patients with treatment resistant depression.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Other: Algorithm guided treatment (AGT) — AGTs consist of strategies (which treatments to use), tactics (how to implement each treatment) and treatment steps (in what order to implement the different treatments). Furthermore, AGTs also define critical decision points during the treatment at which the effects of a certain treatment are assessed and based on this assessment recommend specific treatment revisions according to preset "if-then rules." This is most often done by implementing measurement-based care.
  Arms: Algorithm guided treatment (AGT)
Other: Treatment as usual (TAU) — TAU includes the standard clinical care for patients with TRD as determined by a senior consultant.
  Arms: Treatment as usual (TAU)

SUMMARY:
The trial utilizes a pragmatic, randomized, open label design with two parallel arms. Participants aged 18-65 with a diagnosis of unipolar depressive disorder and without stable remission in the past 12 months are randomized 1:1 to receive either algorithm guided treatment (AGT) or treatment as usual (TAU). The AGT approach incorporates pre-defined treatment steps, critical decision points, and "if-then" rules based on symptom response. It leverages prior treatment history, current symptomatology, and tolerability profiles to personalize the therapeutic sequence and reduce treatment inertia. In contrast, TAU reflects standard clinical practice, where treatment decisions are left to clinician discretion without algorithmic structure. The primary objective of the study is to determine whether AGT leads to a greater reduction in depressive symptoms over a 12-week treatment period, as measured by the 6-item Hamilton Depression Rating Scale (HAMD-6). Secondary objectives include evaluating cognitive and psychosocial functioning, suicide risk, treatment adherence, tolerability, number of medication changes, and long-term outcomes at a 24-week follow-up, providing insights into the longer-term trajectory of TRD management.

DETAILED DESCRIPTION:
The study period consists of 12 weeks in the randomized phase and 12-week extended follow up period during which all participants are monitored and treated at the clinician's discretion. After baseline, study visits are planned at 4, 8, 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of unipolar depressive disorder according to ICD-10 based on documented completion of the Mini International Neuropsychiatric Interview, version 7.0.2 (MINI 7.0.2) at Screening and confirmed by medical records or a healthcare professional.
2. Have not achieved stable remission of depression in 12 months at investigator's clinical assessment.
3. Severity of depression: A score of at least 21 on the self-reported Major Depression Inventory (MDI).
4. Age criteria: Subjects must be at least 18 years old and below 65 at the time of randomization.
5. Signed document of informed consent.
6. The participant is an outpatient.
7. No significant change in medical treatment in the last 4 weeks before screening visit.
8. The patient is pharmacologically treated for depression.

Exclusion Criteria:

1. A diagnosis of dementia.
2. Substance misuse influencing study participation as judged by the investigator.
3. High risk of non-adherence at the investigator's discretion.
4. Not understanding the Danish language as judged by the investigator.
5. Suicidality according to C-SSRS with a positive response to question 4 or 5 within the last three months or upon investigator's discretion.
6. Medical conditions such as cancer, kidney failure, epilepsy, deep brain stimulation device, or other medical conditions interfering with study the outcome and safety as judged by investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale, 6 item version (HAMD-6) | From baseline to end of study (12 weeks)
  The primary outcome measure is the Hamilton Depression Scale, 6 item version (HAMD-6), used as a continuous variable. The primary outcome is the difference in differences (DID) between patients randomized to receive algorithm-guided treatment as compared to treatment as usual, as measured by HAMD-6, based on the mITT population.
  The 6-item version of the Hamilton Depression Rating Scale ranges from 0 to 22, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
HAMD-17 | Up to 24 weeks
  All secondary outcomes are based on the mITT population unless otherwise specified. A Per Protocol (PP) analysis at 12 weeks and at the end of follow-up is performed for all continuous secondary outcomes.
  Difference-in-difference in HAMD-17. The 17-item version of the Hamilton Depression Rating Scale ranges from 0 to 52, with higher scores indicating a worse outcome.
HAMD-6 | Up to 24 weeks
  Difference-in-difference in HAMD-6 for the PP12 and the PP24 population. The 6-item version of the Hamilton Depression Rating Scale ranges from 0 to 22, with higher scores indicating a worse outcome.
UKU | Up to 24 weeks
  Difference in difference in UKU adverse events scale
SCIP | Up to 12 weeks
  Difference-in-difference in Screen for Cognitive Impairment in Psychiatry (SCIP).
  Values range from 0 to 64+, higher scores indicating a better outcome.
FAST | Up to 12 weeks
  Difference-in-difference in the Functioning Assessment Short Test (FAST). Values range from 0 to 72, higher scores indicating a worse outcome).
COBRA | Up to 12 weeks
  Difference in difference in Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA). Values range from 0 to 48, higher scores indicating a worse outcome.
CGI | Up to 12 weeks
  Difference in difference in the Clinical Global Impression Scale (CGI). Values range from 1 to 7, higher scores indicating a worse outcome.
C-SSRS | Up to 12 weeks
  Difference in difference in the Columbia-Suicide Severity Rating Scale (C-SSRS).
  Values range from 1 to 5, higher scores indicating a worse outcome.
Between-groups difference in proportion of responders and remitters in HAMD-6 score | Week 8 and 12
  Responders are defined as subjects with a reduction of at least 50 % in their HAMD-6 scores between baseline and the endpoint of interest. Remitters are defined as subjects with HAMD-6 score below 5 at the endpoint of interest. Both are measured at 8 weeks or at a premature endpoint before last-observation-carried-forward (LOCF) and at 12 weeks or at a premature endpoint before LOCF.
Between-group differences in reason for all cause treatment discontinuation | Up to 24 weeks
  Between-group differences in reason for all cause treatment discontinuation (lack of effect, lack of tolerability, lost to follow-up, or other cause)
Between-group differences in time to all cause treatment discontinuation | Up to 24 weeks
  Between-group differences in time to all cause treatment discontinuation
Between-group differences in number of changes in treatment strategies | Up to 12 weeks
  Between-group differences in number of changes in treatment strategies
Between-group differences in number of changes in the number of different prescribed medications over the treatment period | Up to 12 weeks
  Between-group differences in number of changes in the number of different prescribed medications over the treatment period
Between-group difference for the ITT population in reasons for premature discontinuation | Up to 24 weeks
  Between-group difference for the ITT population in reasons for premature discontinuation
Between-group difference for the ITT population in reasons for time to all cause discontinuation | Up to 24 weeks
  Between-group difference for the ITT population in reasons for time to all cause discontinuation
Between-group difference for the ITT population in adverse events and serious adverse events | Up to 12 weeks
  Between-group difference for the ITT population in adverse events and serious adverse events
Between-groups difference from original randomization in proportion of responders and remitters at end of follow-up | Up to 24 weeks
  Between-groups difference from original randomization in proportion of responders and remitters at end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: René Ernst Nielsen, Prof., MD, PhD, Principal Investigator — Aalborg University Hospital, Psychiatry, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No